CLINICAL TRIAL: NCT02327104
Title: Evaluation of the Effectiveness of the Program of Mindfulness - Based Relapse Prevention (MBRP) as an Assistant Strategy to the Treatment of Tobacco Dependence
Brief Title: Effectiveness of Mindfulness Based Relapse Prevention for Tobacco Dependents
Acronym: MBRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ana Regina Noto, PhD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROCESSO FAPESP 2013/02316-5
Record Dates: First submitted 2014-12-21; First posted 2014-12-30 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Tobacco Use Disorder
Keywords: mindfulness; tobacco dependence; relapse prevention
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Relapse Prevention (Experimental): The Experimental Group (EG) will undergo eight sessions of MBRP after Brazilian Ministry of Health Protocol (BMHP) for Tobacco dependence treatment. MBRP Program: the first three sessions: focus on practicing mindful awareness and integrating mindfulness practices into daily life (body scan, sitting meditation, walking meditation); The next three sessions: emphasize acceptance of present experience and application of mindfulness practices to relapse prevention; The final two sessions: expand to include issues of self-care, support network, and lifestyle balance.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention
- Brazilian Ministry of Health Protocol (Other): The Control Group (CG) is undergo the protocol of the Brazilian Ministry of Health Protocol (BMHP): clinical evaluation, four sessions of cognitive-behavioral approach and Nicotine Replacement Therapy and/or Bupropion as needed, as the Experimental Group. And during the eight sessions of MBRP (EG) both groups (EG and CG) are subjected to eight maintenance sessions of BMHP.
  Interventions: Behavioral: Mindfulness Based Relapse Prevention; Other: Brazilian Ministry of Health Protocol

INTERVENTIONS:
Behavioral: Mindfulness Based Relapse Prevention — The MBRP is an adjuvant treatment for people that have been treated for drug use related problems, and to prevent relapses.
Other: Brazilian Ministry of Health Protocol — The control group will receive maintenance sessions based on the Ministry of Health protocol after the four sessions of cognitive-behavioral approach.
  Arms: Brazilian Ministry of Health Protocol

SUMMARY:
The dependence on tobacco is a predictable leading cause of death. The treatment based on the cognitive-behavioral therapy, including relapse prevention, became standard for tobacco dependents; yet scientific advances are still needed. Accordingly, the Mindfulness-Based Relapse Prevention (MBRP) program, adjunct to treatment, has shown promising results. The purpose of this project is to evaluate the effectiveness of the program MBRP as an adjunct in the treatment of smoking cessation instituted by the Ministry of Health, through the Instituto Nacional do Câncer (INCA) in Brazil.There will be a randomized clinical trial, with a simple random allocation. 60 patients will participate in this study receiving treatment (INCA'S standard) randomized between two groups: the MBRP Group (EG), which will undergo eight sessions of MBRP; and the Control Group (CG) that will undergo eight sessions of the traditional model of Relapse Prevention.This study will be conducted at Ambulatory benchmark to smoking cessation treatment in the city of Juiz de Fora (Minas Gerais State- Brazil). Changes will be evaluated on several variables such as cessation of smoking, anxiety, depression, craving, positive and negative affects and will investigate the association of levels of mindfulness with smoking cessation. The data will be assessed at baseline (T0) and four other times: 1 (T1), 3 (T2), 6 (T3) and 12 months (T4) after the initiation of the study, besides being subjected to evaluations of regularly planned maintenance in the protocol of Ministry of Health. For data analysis there will be used Analysis of Variance with Repeated Measures and Longitudinal Logistic Regression, in order to evaluate the effect of two types of intervention on the evolution of comorbidities and abstinence of patients.

DETAILED DESCRIPTION:
Treatments based on cognitive-behavioral therapy, including relapse prevention, have become standard for smoking cessation in Brazil and many other areas of the world; yet scientific advances are still needed.

Mindfulness-based approaches have more recently begun to be assessed and implemented for treatment of addiction. The Mindfulness-Based Relapse Prevention (MBRP) program, which integrates mindfulness practice with cognitive therapy approaches, has shown promising preliminary results in previous studies.

The purpose of the current study is to evaluate the effectiveness of the Mindfulness-Based Relapse Prevention program as an adjunct in the standard smoking cessation treatment instituted by the Ministry of Health in Brazil.

The study is a randomized clinical trial, with 60 patients diagnosed with nicotine dependence. 60 patients will participate in this study receiving treatment (instituted by the Ministry of Health in Brazil, through the Instituto Nacional do Câncer - INCA'S standard) randomized between two groups: the Experimental Group (EG), which will undergo eight sessions of MBRP; and the Control Group (CG) that will undergo eight sessions of the traditional model of Relapse Prevention (INCA's standard). This will include patients diagnosed with nicotine dependence, who have achieved abstinence. Specific Objetctives: Evaluate the difference in the number of patients who continued abstinence of tobacco; Study the effectiveness MBRP in preventing lapses and relapses; Evaluate the effect of MBRP on the craving and its association with smoking cessation; Evaluate the effect of MBRP in positive and negative affects and its association with smoking cessation; To investigate the association of levels of mindfulness with smoking cessation; Evaluate the effect of MBRP in depressive symptoms, and its possible association with smoking cessation; Evaluate the effect of MBRP in anxiety symptoms, and its possible association with smoking cessation. These will be assessed at baseline (T0) and four other times: 1 (T1), 3 (T2), 6 (T3) and 12 months (T4) after the initiation of the study, besides being subjected to evaluations of regularly planned maintenance in the protocol INCA. Screening instruments: Self Report Questionnaire (SRQ-20); Questionnaire of Smoking Urges (QSU); Hospital Anxiety and Depression Scale (HAD); Center for Epidemiologic Studies Depression Scale (CES-D); Five Facet Mindfulness Questionnaire (FFMQ); Smokerlyser (measuring CO); The Fagerstrom Test for Nicotine Dependence (FTND); Positive and Negative Affect Schedule (PANAS). For data analysis there will be used Analysis of Variance with Repeated Measures and Longitudinal Logistic Regression, in order to evaluate the effect of two types of intervention on the evolution of comorbidities and abstinence of patients. Context: Ambulatory benchmark to smoking cessation treatment in the city of Juiz de Fora, Minas Gerais, Brazil. Participants: • Inclusion: patients with a diagnosis of nicotine dependence;• Exclusion: dependence on other substances, psychiatric comorbidities, pregnant women. •Groups matched for gender, education level and dependence on tobacco level. This initial study will evaluate the feasibility of Mindfulness-Based Relapse Prevention in the context of the Brazilian Public Health system as a supplemental treatment on craving and smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of nicotine dependence;
* Patients currently smoking at least 10 cigarettes a day;
* Do not have any current major psychological disorders;
* Patients undergoing treatment for the first time
* Be willing to attend treatment and follow-up sessions, complete surveys and expired CO tests;
* Do not exhibit dependence on other drugs.

Exclusion Criteria:

* Dependence on other substances;
* Psychiatric comorbidities;
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in the maintenance of abstinence from Cessation of tobacco use through assessment interviews (self-report and CO monitor will be used), and the point prevalence | baseline and twelve months
  We will assess the maintenance of abstinence from tobacco use through assessment interviews (self-report and CO monitor will be used), and the point prevalence will be the primary outcome measure.

SECONDARY OUTCOMES:
Change in smoking urges measured with the self report questionnaire: Questionnaire of Smoking Urges (QSU) | baseline and twelve months
  This will be measured with the self report questionnaire: Questionnaire of Smoking Urges (QSU)
Change in Symptoms of Anxiety measured through the The Hospital Anxiety and Depression Scale (HAD) | baseline and twelve months
  The symptoms of anxiety will be measured through the The Hospital Anxiety and Depression Scale (HAD)
Change in Symptoms of Depression measured through the Centre for Epidemiologic Studies Depression Scale (CES-D) | baseline and twelve months
  The symptoms of depression will be measured through the Centre for Epidemiologic Studies Depression Scale (CES-D)
change in Self report Mindfulness level measured with the self report questionnaire Five Facet Mindfulness Questionnaire (FFMQ) | baseline and twelve months
  This will be measured with the self report questionnaire Five Facet Mindfulness Questionnaire (FFMQ)
Maintenance of Abstinence measured by a Bedfont Micro Smokerlyser - CO monitor | baseline and twelve months.
  Abstinence will be measured by a Bedfont Micro Smokerlyser - CO monitor, to support self-reports of smoking cessation.
Tobacco Dependence measured through The Fagerstrom Test for Nicotine Dependence (FTND) | baseline and twelve months
  This will be measured through The Fagerstrom Test for Nicotine Dependence (FTND)
Change in Positive and Negative Affects measured through Positive and Negative Affect Scale (PANAS) | baseline and twelve months
  This will be measured through Positive and Negative Affect Scale (PANAS).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Regina Noto, Doctor, Study Director — Federal University of São Paulo
Locations (1):
- Drug Dependency Unit of the Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700
- [Derived] Weiss de Souza IC, Kozasa EH, Bowen S, Richter KP, Sartes LMA, Colugnati FAB, Noto AR. Effectiveness of Mindfulness-Based Relapse Prevention Program as an Adjunct to the Standard Treatment for Smoking: A Pragmatic Design Pilot Study. Nicotine Tob Res. 2020 Aug 24;22(9):1605-1613. doi: 10.1093/ntr/ntaa057. PMID 32222767